CLINICAL TRIAL: NCT03136965
Title: Platelet-Rich Plasma (PRP) Therapy for Patellar Tendinopathy: A Randomized Controlled Trial Correlating Clinical, Biomechanical and Novel Imaging Biomarkers
Brief Title: Platelet-Rich Plasma Therapy for Patellar Tendinopathy
Acronym: PRP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: General Electric (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2016-0811; A539300 (Other: UW Madison); SMPH/RADIOLOGY/RADIOLOGY* (Other: UW Madison); Protocol Ver 0.15, 12/23/2021 (Other: UW Madison)
Record Dates: First submitted 2017-04-06; First posted 2017-05-02 (Actual); Results first posted 2023-10-26 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Patellar Tendinitis
MeSH Terms: interventions — Dry Needling

STUDY DESIGN:
Intervention Model Description: Double-blinded randomized controlled trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Subjects and assessors will be blinded to the subject group allocation. Subjects will be identified to study personnel using a unique study number only and results of the imaging studies will be blinded, batched, and evaluated in a randomized manner.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Platelet-Rich Plasma (PRP) (Experimental): Group 1 (PRP) will receive a single US-guided injection of 5 mL autologous PRP.
  Interventions: Biological: PRP
- Dry Needling Procedure (Placebo Comparator): Group 2 (dry needling) will undergo US-guided dry needling procedure similar to PRP injection.
  Interventions: Procedure: Dry Needling
- Sham Procedure (Sham Comparator): Group 3 (sham) will undergo US-guided sham dry needling procedure.
  Interventions: Procedure: Dry Needling - Sham

INTERVENTIONS:
Biological: PRP — Injection of autologous platelet rich plasma (PRP)
  Arms: Platelet-Rich Plasma (PRP)
Procedure: Dry Needling — This is a therapeutic procedure that involves the same injection procedures under ultrasound guidance as in the PRP group but no PRP will be injected inside the patellar tendon.
  Arms: Dry Needling Procedure
Procedure: Dry Needling - Sham — This is a sham procedure that involves similar injection procedures under ultrasound guidance as in the PRP and DN groups with no injection of PRP or needle placement inside the patellar tendon.
  Arms: Sham Procedure

SUMMARY:
The overall goal of this research is to find an effective treatment for patellar tendinopathy (PT). To achieve this, we will conduct a double-blinded randomized controlled trial to investigate if platelet-rich plasma is effective for treatment. Clinical (pain and function scores) and bio-mechanical (knee strength) measures will be correlated with disease modification changes assessed using conventional and novel quantitative magnetic resonance imaging (MRI) and ultrasound (US) techniques.

DETAILED DESCRIPTION:
Sixty-six patients with PT will be randomized to one of three study arms. Subjects in Group 1 (PRP) will receive a single US-guided injection of 5 milliliters of autologous PRP into the patellar tendon, subjects in Group 2 (DN) will undergo ultrasound guided dry needling of the patellar tendon, and subjects in Group 3 (SH) will undergo a sham control ultrasound guided dry needling in the subcutaneous tissue only (not intratendon) at the level of the patellar tendon. The efficacy of the different treatment options will be assessed by pain- and function-dependent, PT-specific Victorian Institute of Sport Assessment Patella (VISA-P) quality of life scores, activity level scores, knee strength measurements, and conventional and novel MRI and US imaging at baseline, 16, 32, and 52 weeks post-treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 39 years
2. Chronic (>3 months) PT
3. Clinical examination consistent with PT
4. MRI or US confirmation of PT
5. Pain score of 3 or greater on a 10-point visual analogue scale
6. Self-report failure of supervised physical therapy
7. Self-report failure of at least 2 of the most common treatment options for PT (e.g. NSAIDs, relative rest, ice and bracing).

Exclusion Criteria:

1. Inability to comply with study follow-up requirements
2. History of bleeding disorders or other hematologic conditions
3. Knee pain from other possible etiologies (e.g., degenerative joint disease, meniscal tear, ligament injury or reconstruction)
4. Full or partial patellar tendon tear
5. Current use of anticoagulation or immunosuppressive therapy
6. Prior knee trauma requiring medical attention or surgery
7. Worker's compensation injury
8. Daily opioid use for pain
9. Contraindication to MRI.
10. Systemic diseases such as Diabetes and connective tissue diseases.
11. Prior PRP or DN procedure.
12. Women that are pregnant

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2017-04-25 (Actual); Primary Completion 2022-08-15 (Actual); Study Completion 2022-08-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Lee, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from April 2017 to June 2021.
Pre-assignment Details: One person was consented and enrolled to the study, but post-imaging analysis, did not have patellar tendinopathy and did not fully onboard to study.
Period: Overall Study
Arm/Group | Platelet-Rich Plasma (PRP) | Dry Needling Procedure | Sham Procedure
Started | 10 | 10 | 9
Completed | 10 | 9 | 9
Not Completed | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Platelet-Rich Plasma (PRP) | Dry Needling Procedure | Sham Procedure | Total
Number analyzed (Participants) | 10 | 10 | 9 | 29
Age, Customized [Count of Participants; unit: Participants]
  20-29 years old | 7 | 6 | 7 | 20
  30-39 years old | 3 | 4 | 2 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 2 | 5
  Male | 9 | 8 | 7 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 9 | 10 | 8 | 27
  Unknown or Not Reported | 1 | 0 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 8 | 10 | 6 | 24
  More than one race | 1 | 0 | 0 | 1
  Unknown or Not Reported | 1 | 0 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 9 | 29

OUTCOME MEASURES:

1. Primary Outcome: Change in Measure of Pain Level: VISA-P Score
Description: A quality of life measure, the Victoria Institute of Sport Assessment - Patellar Tendon (VISA-P) will be used to evaluate pain before and after the intervention. The instrument is scored from 0-100 with higher scores indicating less pain.
Time Frame: baseline, 16 weeks, 32 weeks, 52 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Platelet-Rich Plasma (PRP) | Dry Needling Procedure | Sham Procedure
Number analyzed (Participants) | 10 | 10 | 9
score on a scale
  baseline | 32.2 (57.8) | 46.3 (69.5) | 43.2 (68.8)
  16 weeks | 52.5 (78.1) | 56.9 (82) | 53.7 (79.4)
  32 weeks | 62.1 (87.7) | 56.2 (81.3) | 58.9 (85.7)
  52 weeks | 64 (89.6) | 55.6 (83) | 60.3 (87)

2. Primary Outcome: Change in Measure of Activity Level: Tegner Activity Level Score
Description: The Tegner Activity Level Score will be used to evaluate activity level before and after the intervention. It is scored from 0-10 with 0 indicating disability and 10 competitive elite sport.
Time Frame: baseline, 16 weeks, 32 weeks, 52 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Platelet-Rich Plasma (PRP) | Dry Needling Procedure | Sham Procedure
Number analyzed (Participants) | 10 | 10 | 9
score on a scale
  baseline | 2.8 (5.2) | 5 (7.2) | 5.3 (7.8)
  16 weeks | 3.5 (6) | 4.5 (6.9) | 4.6 (7.1)
  32 weeks | 4.2 (6.7) | 5.1 (7.5) | 4.5 (7)
  52 weeks | 4.8 (7.3) | 5.2 (7.9) | 4.5 (7)

3. Primary Outcome: Change in Visual Analogue Scale (VAS) Pain Score
Description: Participant pain level was assessed using a VAS score from 0 (no pain) to 10 (worst pain).
Time Frame: baseline, 16 weeks, 32 weeks, 52 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Platelet-Rich Plasma (PRP) | Dry Needling Procedure | Sham Procedure
Number analyzed (Participants) | 10 | 10 | 9
score on a scale
  baseline | 5.9 (9) | 5.5 (8.3) | 6.1 (9.2)
  16 weeks | 2.5 (5.6) | 4.2 (7.2) | 2.9 (6)
  32 weeks | 1.1 (4.1) | 3.8 (6.8) | 1.6 (4.7)
  52 weeks | 0 (3.2) | 2.8 (6.1) | 1.8 (4.9)

4. Secondary Outcome: MRI Scan To Demonstrate Treatment-related Changes in Pathologic Imaging Features of PT (T2 Signal Intensity)
Description: To demonstrate treatment-related changes in pathologic imaging features of PT using conventional MRI measures.
Time Frame: baseline, 16 weeks, 52 weeks
Population: T2 signal intensity was not measured via MRI, rather MRI was used for exploratory measures using novel software as updated in the Other Pre-specified measures.
Arm/Group | Platelet-Rich Plasma (PRP) | Dry Needling Procedure | Sham Procedure
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: MRI Scan To Demonstrate Treatment-related Changes in Pathologic Imaging Features of PT (Thickness)
Description: To demonstrate treatment-related changes in pathologic imaging features of PT using conventional MRI measures.
Time Frame: baseline, 16 weeks, 52 weeks
Population: MRI was not used to measure thickness, Ultrasound was used to assess thickness.
Arm/Group | Platelet-Rich Plasma (PRP) | Dry Needling Procedure | Sham Procedure
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Ultrasound Scan to Demonstrate Treatment-related Changes in Pathologic Imaging Features of PT (Thickness)
Description: To demonstrate treatment-related changes in pathologic imaging features of PT using conventional ultrasound measures.
Time Frame: baseline, 16 weeks, 52 weeks
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Platelet-Rich Plasma (PRP) | Dry Needling Procedure | Sham Procedure
Number analyzed (Participants) | 10 | 10 | 9
millimeters
  baseline | 6.6 (8.6) | 5.2 (7.1) | 7 (9)
  16 weeks | 6.5 (8.5) | 5.4 (7.3) | 7 (9.1)
  52 weeks | 6 (8) | 5.4 (7.4) | 5.7 (7.7)

7. Secondary Outcome: Ultrasound Scan to Demonstrate Treatment-related Changes in Pathologic Imaging Features of PT (Echogenicity) From Baseline
Description: To demonstrate treatment-related changes in pathologic imaging features of PT using conventional ultrasound measures. Echogenicity is the grey scale images found on standard B-mode exams. The grey scale can change with pathology, therefore, the grading scale is implemented. The data reported are scores from a grading system, where 0 - normal; 1- mild; 2- moderate; 3- severe.
Time Frame: baseline, 16 weeks, 52 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Platelet-Rich Plasma (PRP) | Dry Needling Procedure | Sham Procedure
Number analyzed (Participants) | 10 | 10 | 9
score on a scale
  baseline | 1.3 (2.5) | 1.5 (2.5) | 1.4 (2.6)
  Change from Baseline at 16 weeks | 1.3 (2.5) | 1.3 (2.4) | 1.9 (3)
  Change from Baseline at 52 weeks | 1.3 (2.5) | 1.4 (2.6) | 1.1 (2.3)

8. Secondary Outcome: Ultrasound Scan to Demonstrate Treatment-related Changes in Pathologic Imaging Features of PT (Hyperemia) From Baseline
Description: To demonstrate treatment-related changes in pathologic imaging features of PT using conventional ultrasound measures. Hyperemia means an increase in the number of blood vessels, it is scored on a semi-qualitative scale where 0 - normal; 1- mild; 2- moderate; 3- severe. If there's an improvement in hyperemia grading then the score decreases.
Time Frame: baseline, 16 weeks, 52 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Platelet-Rich Plasma (PRP) | Dry Needling Procedure | Sham Procedure
Number analyzed (Participants) | 10 | 10 | 9
score on a scale
  baseline | 1.1 (2.5) | 0.6 (1.8) | 1.4 (2.8)
  Change from Baseline at 16 weeks | 0.7 (2) | 0.4 (1.7) | 1.3 (2.7)
  Change from Baseline at 52 weeks | 0.4 (1.8) | -0.2 (1.2) | 0.4 (1.8)

9. Other Pre Specified Outcome: Isokinetic Dynamometer Measure of Flexor and Extensor Muscle Strength Before and After the Intervention
Description: Flexor and extensor muscle strength will be measured with this device before and after the intervention.
Time Frame: baseline, 16 weeks, 52 weeks
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Relationship Between Changes in Novel Quantitative MRI and US Parameters of PT and Clinical and Biomechanical Improvement Following Treatment.
Description: To investigate the relationship between changes in novel quantitative MRI techniques and US parameters of PT and clinical and biomechanical improvement following treatment.
Time Frame: 52 weeks
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Ultrashort Time to Echo (UTE) T2* Relaxation Time (T2*Single)
Description: Exploratory MRI measure
Time Frame: baseline, 16 weeks, 52 weeks
Reporting Status: Not Posted

12. Other Pre Specified Outcome: T2* Fraction of Fast-relaxing Macromolecular-bound Water (FF)
Time Frame: baseline, 16 weeks, 52 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: up to 52 weeks
Arm/Group | Platelet-Rich Plasma (PRP) | Dry Needling Procedure | Sham Procedure
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/9
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-23): https://cdn.clinicaltrials.gov/large-docs/65/NCT03136965/Prot_SAP_000.pdf